CLINICAL TRIAL: NCT03065387
Title: Phase I Study of the Pan-ERBB Inhibitor Neratinib Given in Combination With Everolimus, Palbociclib, or Trametinib in Advanced Cancer Subjects With EGFR Mutation/Amplification, HER2 Mutation/Amplification, or HER3/4 Mutation or KRAS Mutation
Brief Title: Neratinib and Everolimus, Palbociclib, or Trametinib in Treating Participants With Refractory and Advanced or Metastatic Solid Tumors With EGFR Mutation/Amplification, HER2 Mutation/Amplification, or HER3/4 Mutation or KRAS Mutation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0430; NCI-2018-01218 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0430 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; EGFR Gene Amplification; EGFR Gene Mutation; ERBB2 Gene Amplification; ERBB2 Gene Mutation; ERBB3 Gene Mutation; ERBB4 Gene Mutation; KRAS Gene Mutation; Metastatic Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Everolimus; neratinib; palbociclib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (neratinib, everolimus) (Experimental): Participants receive neratinib PO daily and everolimus PO daily. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Drug: Neratinib
- Arm II (neratinib, palbociclib) (Experimental): Participants receive Neratinib PO daily for 28 days and Palbociclib PO daily for 21 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Neratinib; Drug: Palbociclib
- Arm III (neratinib, trametinib) (Experimental): Participants receive neratinib PO daily and trametinib PO daily as directed. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Neratinib; Drug: Trametinib

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
  Arms: Arm I (neratinib, everolimus)
Drug: Neratinib — Given PO
  Other Names: (2E)-N-(4-((3-chloro-4-((pyridin-2-yl)methoxy)phenyl)amino)-3-cyano-7-ethoxyquinolin-6-yl)-4-(dimethylamino)but-2-enamide; HKI 272; HKI-272; PB 272; PB-272
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991
  Arms: Arm II (neratinib, palbociclib)
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist
  Arms: Arm III (neratinib, trametinib)

SUMMARY:
This phase I trial studies the side effects and best dose of neratinib in combination with everolimus, palbociclib, or trametinib in participants with solid tumors with EGFR mutation/amplification, HER2 mutation/amplification, HER3/4 mutation, or KRAS mutation that do not respond to treatment (refractory) and have spread to other parts of the body (advanced or metastatic). Neratinib, palbociclib, and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as everolimus, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving neratinib with everolimus, palbociclib, or trametinib may work better than neratinib alone in treating participants with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of neratinib when combined with one of the following agents:

Ia. Arm 1: Everolimus (mTOR inhibitor) Ib. Arm 2: Palbociclib (CDK 4/6 inhibitor) Ic. Arm 3: Trametinib (MEK inhibitor). II. To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of neratinib combination therapy.

SECONDARY OBJECTIVES:

I. To determine preliminary anti-tumor efficacy of neratinib combination therapy.

II. To determine pharmacodynamic markers in tissue, blood and plasma that may predict outcome.

III. To explore the potential of drug-drug interactions by evaluating the pharmacokinetic profile of each agent when administered in these combinations: neratinib+everolimus, neratinib+palbocclib, and neratinib+trametinib and blood-based biomarkers.

EXPLORATORY OBJECTIVES:

I. To determine baseline molecular markers (deoxyribonucleic acid [DNA], ribonucleic acid [RNA] and protein) that may predict clinical benefit.

II. To determine concordance of human epidermal growth factor receptor mutation (EGFR, HER2, HER3, and HER4) or EGFR, HER2 amplification in archival tissue and pre-treatment biopsies. Impact of these correlatives on response will be explored.

III. To determine concordance of human epidermal growth factor receptor mutation (EGFR, HER2, HER3, and HER4) or EGFR, HER2 amplification in tumor and cell-free DNA (cfDNA). Impact of these correlatives on response will be explored.

IV. To utilize cfDNA from plasma specimens collected during the course of treatment to explore mechanisms of primary and acquired resistance to neratinib combination therapy.

OUTLINE: This is a dose-escalation study. Participants are assigned to 1 of 3 arms.

ARM I: Participants receive neratinib orally (PO) daily and everolimus PO daily. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Participants receive neratinib PO daily and palbociclib PO daily for 3 weeks followed by 1 week off. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM III: Participants receive neratinib PO daily and trametinib PO daily as directed. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with advanced or metastatic solid tumors that are refractory to standard therapies known to provide clinical benefit. Subjects with hematologic malignancy including lymphoma/myeloma will not be enrolled on this study.
2. Subjects must have one of the following:

   1. somatic mutations in human epidermal growth factor receptor (EGFR, HER2, HER3, and HER4)
   2. EGFR gene amplification (patients with 3+ results on immunohistochemistry testing for EGFR may be allowed to enroll if gene amplification results are unavailable)
   3. HER2 gene amplification (patients with 3+ results on immunohistochemistry testing for Her-2 may be allowed to enroll if gene amplification results are unavailable)
   4. Somatic mutation in KRAS (Patients will be enrolled only on neratinib and trametinib combination ARM).
3. Subjects must have measurable disease by RECIST v1.1. (only for MTD Expansion Cohorts)
4. Subjects must be ≥18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
6. Abnormal organ function is permitted. However, subjects must have:

   1. absolute neutrophil count ≥ 1500/mL
   2. platelets ≥ 100,000/mL
   3. hemoglobin ≥ 9 g/dL
   4. creatinine ≤ 1.5 X upper limit of normal (ULN) or CrCl >40 ml/min
   5. total bilirubin ≤ 1.5 X ULN
   6. aspartate aminotransferase (AST/SGOT) and/or alanine aminotransferase (ALT/SGPT) ≤ 2.5 X ULN (≤5 X ULN in subjects with liver metastases)
7. Subjects must be ≥4 weeks or at least 5 half-lives beyond treatment with any chemotherapy or other investigational therapy to include hormonal, biological, or targeted agents, whichever is shorter at the time of treatment initiation. Subjects must be ≥4 weeks beyond treatment with wide field radiation therapy or ≥2 weeks for limited field radiation therapy for palliation (not including whole brain radiation or stereotactic radiotherapy, for which subjects must be ≥4 weeks beyond treatment).
8. Women of child-bearing potential MUST have a negative serum or urine human chorionic gonadotropin (HCG) test unless prior hysterectomy or menopause (defined as 12 consecutive months of amenorrhea). Subjects should not become pregnant or breastfeed while on this study. Sexually active subjects must agree to use contraception for the duration of study participation and for 4 months after the last dose of neratinib and everolimus, palbociclib or trametinib.
9. Ability to understand and willingness to sign informed consent form prior to initiation of the study and any study procedures.

   Only for subjects enrolled in Arm 1 - Neratinib and Everolimus
10. Fasting lipid profile: Cholesterol less than or equal to 350 mg/dL and triglycerides less than or equal to 400 mg/dL.
11. Subjects who are taking medications with potent inhibitors or inducers of CYP450 3A4 should be off for 5 half-lives prior to starting everolimus.

    Only for subjects enrolled in Arm 2 - Neratinib and Palcociclib
12. Any prior neuropathy should be back to baseline or grade 1
13. Subjects who are taking medications with potent inhibitors or inducers of CYP450 3A4 should be off for 5 half-lives prior to starting Palbociclib.

    Only for subjects enrolled in Arm 3 - Neratinib and Trametinib
14. All skin rash (dermatitis acneiform, erythema, xeroderma, eczema) should be at grade 1 when starting trametinib treatment.
15. History of retinal disorder, dry eye syndrome, or blurry vision need to be evaluated by ophthalmology prior to starting treatment.

Exclusion Criteria:

1. Subjects who are pregnant or breastfeeding;
2. Known Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV) infection.
3. Inability or unwillingness to swallow pills.
4. Active infection requiring intravenous (IV) antibiotics or other uncontrolled intercurrent illness requiring hospitalization.
5. Clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels. For example, subjects should have no more than 50% of the large intestine removed and no sign of malabsorption (e.g. gastrectomy, ileal bypass, chronic diarrhea, Crohn's disease, malabsorption, gastroparesis).
6. Inability to comply with the study and follow-up procedures.
7. History of cerebrovascular accident (CVA), myocardial infarction or unstable angina within the previous 6 months before starting therapy.
8. Prolongation of QT/QTc interval (QTc interval >450 ms for males or >470 ms for females) using the Fredericia method of QTc analysis. For patients with bundle branch block (BBB), the Rautaharju method of QTc analysis (QTcR) will be used.
9. Has active primary brain tumor, active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks with no neurological symptoms, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless or clinical stability.
10. Uncontrolled concurrent disease or illness including but not limited to:

    * symptomatic congestive heart failure (NYHA Class III or IV) per the NYHA Classification (see Appendix B), unstable angina pectoris, clinically significant cardiac arrhythmia
    * unstable or untreated cardiac conditions or ejection fraction of <50% as determined by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA)
    * diabetes mellitus (i.e. fasting blood glucose >220 despite acceptable chronic diabetes therapy)
    * psychiatric illness that would limit compliance with study requirements, as determined by the investigator
11. Participating in any other clinical trials using an investigational product. Only for subjects enrolled in Arm 1 - Neratinib and Everolimus
12. History of hypersensitivity to everolimus
13. Subjects requiring therapy with immunosuppressive agents such as anti-tumor necrosis factor alpha (TNFα) agents (Etanercept, Adalimumab), azathioprine, methotrexate, cyclosporine, etc for active autoimmune disorder.
14. Major surgery ≤28 days prior to treatment with everolimus. Only for subjects enrolled in Arm 3 - Neratinib and Trametinib
15. Albumin less than 3 Gm/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of neratinib when given in combination with everolimus, palbociclib, or trametinib | Up to 28 days
  Defined by dose-limiting toxicity (DLT). The MTD will be defined as the highest dose at which no more than 1 of 6 evaluable subjects has had a DLT.

SECONDARY OUTCOMES:
Incidence of adverse events of neratinib when given in combination with everolimus, palbociclib, or trametinib | Up to 30 days post last dose
  National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 will be used to quantify the intensity of adverse events occurring during treatment in this study.
Objective response | Up to 5 years
  Per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The anti-tumor efficacy of each combination will be evaluated by objective response by RECIST v1.1. This analysis will not utilize statistical analysis per standard phase I trials.
Determination of pharmacodynamics markers in tissue, blood, and plasma | Up to completion of treatment
  Pharmacodynamics markers in tissue, blood, and plasma will be determined that may predict outcome and exploration of the pharmacokinetic profile of each agent when administered in combination. Marker values will be compared between subjects with and without clinical benefit using chi-squared or Fisher exact tests for categorically-scaled markers and Wilcoxon rank sum tests for interval- and ordinal-scaled markers. Due to the large number of candidate markers, only those significant on univariate analysis will be combined into a single logistic regression model to assess their independent effects on clinical benefit. Analyses will be performed both within and across the three cohorts. Results will be considered exploratory and thus no corrections will be made for multiple testing.

CONTACTS AND LOCATIONS:
Overall Officials: Sarina A Piha-Paul, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Piha-Paul SA, Tseng C, Tran HT, Gao M, Karp DD, Subbiah V, Tsimberidou AM, Kawedia JD, Fu S, Pant S, Yap TA, Morris VK, Kee BK, Blum Murphy M, Lim J, Meric-Bernstam F. A phase I trial of the pan-ERBB inhibitor neratinib combined with the MEK inhibitor trametinib in patients with advanced cancer with EGFR mutation/amplification, HER2 mutation/amplification, HER3/4 mutation or KRAS mutation. Cancer Chemother Pharmacol. 2023 Aug;92(2):107-118. doi: 10.1007/s00280-023-04545-4. Epub 2023 Jun 14. PMID 37314501
- See also: MD Anderson Cancer Center — http://www.mdanderson.org